CLINICAL TRIAL: NCT05525598
Title: Internet-based Treatment for Patients Suffering From Severe Functional Somatic Disorders: A Randomized Controlled Trial.
Brief Title: Internet-based Treatment for Patients Suffering From Severe Functional Somatic Disorders
Acronym: OneSTEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Sygehus Lillebaelt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OneStep v2.0
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Bodily Distress Disorder Moderate; Bodily Distress Disorder Severe; Fibromyalgia; Chronic Fatigue Syndrome; Irritable Bowel Syndrome; Somatization
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-delivered therapist-assisted treatment: "One step at the time" (Experimental): "One step at the times" consists of 11 internet-delivered modules delivered over 14 weeks. Each module explores a different theme, primarily including elements from Cognitive Behavioral Therapy (CBT) for FSD, and includes FSD-related psychoeducation, various interactive exercises, and video and audio material. Interactions between patients and the therapist will take place via the telephone 3 times (start, mid-term, and end-of-treatment) and embedded messaging (therapist will respond to patients) approx. 2 times a week. The participating therapists are supervised every other week by specialized psychologists.
  Interventions: Behavioral: "One step at a time"
- Internet-delivered non-guided treatment: "Get started" (Active Comparator): "Get started" is a non-guided self-help program, developed as an active control, that includes 4 modules consisting of FSD-related psychoeducation and guidance on making lifestyle improvements. Participants will have access to the "Get started" program for 14 weeks.
  Interventions: Behavioral: "Get started"

INTERVENTIONS:
Behavioral: "One step at a time" — [see 'arms' section for full description]
  Arms: Internet-delivered therapist-assisted treatment: "One step at the time"
Behavioral: "Get started" — [see 'arms' section for full description]
  Arms: Internet-delivered non-guided treatment: "Get started"

SUMMARY:
The aim of this multi-center, two-armed, randomized controlled trial is to assess the effect of a novel internet-based therapist-assisted treatment program "One step at a time" designed for the treatment of patients with moderate to severe functional somatic disorder (FSD).

The trial will enroll 166 patients with FSD who will be randomized (1:1) to either the experimental condition (14 weeks' treatment with "One step at a time") or the active control condition ("GetStarted"), which is a non-guided internet-based treatment program for patients with FSD. The trial will include patients aged 18-60 years with an established single/oligo-organ or multi-organ FSD diagnosis, with a duration of minimum 6 months. The primary outcome measures will be based on self-reported physical health (SF-36 PPH) and treatment satisfaction (CGI-I). The trial will be considered effective if a higher proportion of patients in the experimental condition report a clinically significant outcome compared with patients in the active control condition at the 3-month follow-up after treatment.

DETAILED DESCRIPTION:
OBJECTIVE: To assess the clinical efficacy of the therapist-guided internet-delivered treatment program "One step at a time" for functional somatic disorders (FSDs) compared with an active control "Get Started".

DESIGN: The trial will employ a two-armed randomized, controlled design with an active control condition.

PARTICIPANTS: We will include adult patients (18-60 years) with a medical diagnosis of functional somatic disorder. For a description of eligibility criteria, see the section "Eligibility".

PROJECT GROUP: Thomas Tandrup Lamm (Psychologist, MSc.); Lisbeth Frostholm (Professor, Psychologist, MSc., Ph.D.); Heidi Frølund Pedersen (Associate Professor, Psychologist, MSc., Ph.D.); and Brjánn Ljótsson (Associate Professor, Psychologist MSc., Ph.D.).

The trial will be conducted by the research group at the Dept. of Functional Disorders (www.functionaldisorders.dk), based at Aarhus University Hospital, Denmark. The clinic was established in 1999 and offers assessment and specialized treatment to patients with severe FSD.

The Pain and Headache Clinic (PHC) based at Aarhus University Hospital and the Center for Functional Disorders (CFD) based at Sygehus Lillebælt in Southern Region Denmark will take part in the assessment and recruitment of the patients. The treatment will be conducted by trained therapists, at the Dept. of Functional Disorders.

MAIN HYPOTHESIS: We hypothesize that a statistically significant higher proportion of patients receiving "One-step" will report a clinically relevant improvement in self-reported physical health and self-reported overall health (SF-36 PPH; CGI-I) compared with "Get Started" 3 months after end-of-treatment. Secondarily, that "One step" will be superior to "Get Started" in terms of increasing helpful illness perceptions (IPQ) and behaviors (BRIQ) and reducing illness worry (WI-6-R) 3 months after end-of-treatment.

INTERVENTION: "One step at a time" consists of 11 internet-delivered modules delivered over 14 weeks. The modules are based on previous treatment manuals for group-based psychoeducation and treatment for severe FSD.

The treatment program is developed as a therapist-assisted interactive treatment program. Each module has a specific theme and contains on average between 7 and 10 pages with elements such as psychoeducation; videos of former patients sharing their narrative and treatment experiences; videos of health professionals talking about FSD, symptom understanding, and illness behavior; interactive exercises, graded exercise and exposure, and videos of guided physical stretching and mindfulness exercises.

The modules concerning sleep, diet, and exercise will also be included as additional resources that can be accessed on an-as-needed basis.

The treatment is assisted by a therapist with the purpose of motivating the patient to engage with the treatment, answer questions, and provide assistance with exercises. The interaction is primarily written communication and takes place in an embedded secured message system on the platform. The therapist writes to the patient 1-2 times on a weekly basis. Furthermore, patients are offered 3 supportive telephone consultations during the treatment: 1) A start-up conversation within the first 2 weeks of the treatment, 2) a conversation after module 5 focusing on what the patient has learned so far and what he/she wishes to focus on in the remaining treatment period, and finally 3) an end-of-treatment conversation focusing on how the patient can proceed with those treatment elements from the program that have been most useful. Finally, a module for relatives consisting of videos with health professionals and relatives to patients with severe FSD has been developed.

Treatment is considered completed if the patient has worked actively (logged into the module and completed at least one interactive exercise) in each of the first 5 modules of the treatment program. This was chosen because the enrolled patients will have received the fundamental treatment elements including psychoeducation and an introduction to graded exercise and exposure at this point. The participating therapists are supervised weekly by specialized psychologists with focus on the written interaction in the program.

"Get started" is an internet-delivered non-guided self-help program consisting of 4 brief modules based on pamphlets developed at the Dept of Functional Disorders addressing psychoeducation in severe FSD and a better balance in basic needs like sleep, diet, and exercise. The modules consist of psychoeducation provided by texts giving specific advice on how to improve sleep quality and diet and increase physical activity by applying graded exercise. Participants are encouraged to focus on either sleep, diet, or exercise during the 14-week treatment period.

MEASUREMENTS: Self-reported measures will be administered to both groups at several timepoints during the course of treatment, including before assessment (-2 weeks), before the start of the program (baseline, 0 weeks), after treatment (14 weeks), at the 3-month follow-up (26 weeks, primary endpoint) and at the 12-month follow-up (62 weeks). Beyond this, a smaller selection of process and outcome measures will be administered at weeks 3, 6, and 9. Participants will answer a short list of questions after the completion of each module.

Furthermore, medical doctors will evaluate patients' eligibility and motivation after the initial diagnostic assessment, and after the post-treatment consultation after the 3 month follow-up. Therapists will record number and time usage of telephone consultations throughout the treatment. Both treatment program will continually log the participants' data during the treatment period.

For a detailed list of the measures and measurement time points included, see the section "Outcome measures".

POWER CALCULATION: The power calculation for SF-36 PPH is based on the proportion of patients experiencing a minimum of a 4-point increase in the aggregate score (PPH) from baseline to the 3-month follow-up, which may be regarded as a clinically relevant change (Norman, 2003) and has been used as an indicator of a clinically relevant response to treatment in patients with severe FSD (Schröder et al., 2012; Pedersen et al., 2018).

Based on previous studies, we estimate the proportion experiencing a minimum of a four-point improvement at the primary outcome, PPH to be between 35%-50% in the intervention group and 10-25% in the active control group (Schröder et al., 2012; Fjorback et al., 2013; Pedersen et al., 2018; Pedersen et al., 2019). With a total sample size of N=150 and a proportion in the control group equal to 15%, we will with a power of 81.4% be able to establish a difference between groups if the proportion in the intervention group is a minimum of 35%.

For the CGI-I, patients grade their health as "much worse", "worse", "unchanged", "better", "or much better". In the analyses we collapse "much worse" and "worse" into one category, and "better" and "much better" to one category, which gives us 3 outcomes in each category (worse, unchanged, better). The power analysis is based on an analysis of a proportional odds model with 5% significance level, and 75 patients in the intervention group and 75 persons in the control group. At OR = 2.5 the power will be 79.1%.

We expected an attrition rate of 10% in both groups. Therefore, we chose to include 15 patients beyond the 150 needed. In order to achieve equal group size, we added one more patient. Thus, we aim to include 166 patients in the trial.

ANALYSIS: "Intention to treat" analyses and "completer analysis" will be performed. Directed acyclic graphs will be used to determine the appropriate variables to adjust for. "Completers" are defined as patients who have accessed all of the first 5 modules. A priori hypotheses will be analyzed using logistic regression, mediation analysis (simplex cross-lagged as well as latent growth curve models), and multiple regression. For main analyses single/oligo- and multi-organ BDS patients will be combined and analyzed as an aggregated cohort. We will supplement this with sensitivity analyses, where it will be tested whether FSD type (single/oligo or multi organ) moderates effects. An in-house statistician will be continuously involved in the project.

ETHICAL CONSIDERATIONS: The trial presents low risks (side-effects and/or disadvantages) for the patients who may end their participation at any time point and can get into contact with a physician if their physical/mental health state deteriorates significantly. After patients have reached their final end-point, at the 3-month follow-up, they will be invited to a follow-up consultation with a medical doctor where their health/mental status will be assessed, and the need for further treatment discussed.

A study protocol has been approved by the Research Ethics Board of Aarhus University Hospital for approval (case.nr. 1-10-72-361-21). A pre-registration of the trial has been submitted to ClinicalTrials.gov before the onset of the trial. Data will be handled according to Danish law on the Data Protection Act and the Data Protection Regulation, and have been approved by the Danish Data Protection Agency (case.nr. 772917).

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfil the criteria for moderate-severe FSD operationalized as being diagnosed with either single/oligo-organ BDS, with 2 organ systems that are each affected by 3 or more symptoms, or multi-organ BDS, with 3 or 4 organ systems that are each affected by 3 or more symptoms.
* Patients must have symptom duration > 6 months.
* If older than 25, patients must have been active in the labor market or educational system for at least 12 months during the last 2 years.
* Patient must have access to a computer or tablet with internet connection.
* Patient must be able to understand, read, and write Danish fluently.

Exclusion Criteria:

* Patients are excluded from participation if they present with severe comorbid somatic or psychiatric disease that is insufficiently treated at the time of assessment and is deemed to constitute a potential barrier for engaging in the treatment.
* Patients are excluded if they lack motivation to engage in internet-delivered treatment.
* Patients are excluded if they have poor self-reported IT skills.
* Patients are excluded if they lack informed consent.
* Patients are excluded if they have ongoing treatments with opioids and benzodiazepines.
* Patient's use of psychoactive medications should be stable.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in SF-36 physical health (SF-36 PPH scales) | Pre-assessment (-2 weeks), baseline (0 weeks), during treatment (weeks 3, 6, and 9), after treatment (14 weeks), at 3-month follow up (26 weeks), and at 12-month follow up (62 weeks)
  The SF-36 is a self-reported physical, mental, and social health. Analysis of primary outcome will be based on the PPH subscales. The change that is used to test the main hypothesis is the change from baseline (0 weeks) to 3-month follow-up (26 weeks).
  The full SF-36 is measured at the following time-points: Pre-assessment (-2 weeks), baseline (0 weeks), after treatment (14 weeks), at 3-month follow up (26 weeks), and at 12-month follow up (62 weeks).
  During During treatment (week 3, 6, 9), only the SF-36 PPH subscales (Bodily pain, physical functioning, vitality) will be measured.
Clinical Global Improvement Scale (CGI) | 3-month follow up (26 weeks)
  Single item 5-point self-reported evaluation of overall health improvement. The time point that is used to test the main hypothesis at 3-month follow-up (26 weeks).
  The CGI is measured on the following time points: After treatment (14 weeks), at 3-month follow up (26 weeks), at 12-month follow up (62 weeks)

SECONDARY OUTCOMES:
The Numeric Rating Scale (NRS) | Pre-assessment (-2 weeks), Baseline (0 weeks), During treatment (weeks 3, 6, and 9), After treatment (14 weeks), and at 3 month follow up (26 weeks) at 12 month follow up (62 weeks)
  Self-reported symptom intensity and symptom interference
Emotional distress, anxiety, depression subscales of the 92-item Danish version of the Symptom Checklist (SCL-92) | Pre-assessment (-2 weeks), Baseline (0 weeks), after treatment (14 weeks), at 3-month follow up (26 weeks), and at 12 month follow up (62 weeks).
  Self-reported symptoms of anxiety, depression, and emotional distress
The BDS Checklist-25 | Pre-assessment (-2 weeks), Baseline (0 weeks), after treatment (14 weeks) at 3 month follow up (26 weeks) and at 12 month follow up (62 weeks).
  Self-reported physical symptoms
Whiteley-6 revised | Pre-assessment (-2 weeks), baseline (0 weeks), after treatment (14 weeks), at 3-month follow up (26 weeks), and at 12-month follow up (62 weeks)
  Self-reported illness worries
Brief Illness perception questionnaire (b-IPQ) | Pre-assessment (-2 weeks), Baseline (0 weeks), during treatment (weeks 3, 6, and 9), After treatment (14 weeks), at 3 month follow up (26 weeks) and at 12 month follow up (62 weeks)
  Self-reported illness perceptions
The Behavioural Responses to Illness Questionnaire (BRIQ) | Pre-assessment (-2 weeks), baseline (0 weeks), during treatment (week 3, 6, and 9), after treatment (14 weeks), at 3-month follow up (26 weeks), and at 12-month follow up (62 weeks)
  Self-reported illness behaviour
The credibility/expectancy questionnaire (CEQ) | Before treatment (0 weeks) and after treatment (14 weeks)
  Treatment expectancy, rationale credibility, and treatment satisfaction
Costs associated with Psychiatric Illness (TiC-P) | Before treatment (0 weeks), at 3 month follow up (26 weeks) and at 12 month follow up (62 weeks)
  Self-reported work performance and work absence
The inventory for the assessment of negative effects of psychotherapy (INEP) | After treatment (14 weeks)
  Self-reported negative effects of psychotherapy
The Sources of Meaning and Meaning in Life Questionnaire (SoMe short version) | Baseline (0 weeks), After treatment (14 weeks)
  Self-reported sense of meaningfulness and crisis of meaning
The Internet Evaluation and Utility Questionnaire (iEUQ) | After treatment (14 weeks)
  Self-reported evaluation of the utility of internet-based treatment
Experiences of satisfaction Questionnaire (ESQ) | After treatment (14 weeks)
  Self-reported Patient treatment satisfaction with treatment
Motivation and alliance with therapist (WAI-SR) | Mid-treatment (6 weeks)
  Self-reported experience of therapeutic alliance with therapist
Interoceptive awareness and Sensitivity Questionnaire (ISAQ) | Baseline (0 weeks), After treatment (14 weeks)
  Self-reported tendencies to experience interoception in a neutral or negative way
Emotional Approach Coping scale (EACS) | Baseline (0 weeks), After treatment (14 weeks)
  Self-reported measure of individuals tendency to cope with emotional experiences
Toronto Alexithymia Scale (TAS-20) subscales | Baseline (0 weeks), after treatment (14 weeks)
  Self-reported measure of alexithymia, subscales: Difficulty describing emotions (5 items), Difficulty identifying emotions (7 items)
Experiences in close relations (ECR) | Baseline (0 weeks)
  Self-reported measure of attachment style
Amsterdam Resting State Questionnaire (ARSQ) | Baseline (0 weeks), after treatment (14 weeks), at 3-month follow up (26 weeks)
  Self-reported experiences after short (3 min) resting state exercise.
Somatization sub-scale of the 92-item version of the Symptom Checklist (SCL-92_SOM) | Pre-assessment (-2 weeks), baseline (0 weeks), after treatment (14 weeks) and at 3-month follow up (26 weeks)
  Self-reported somatic symptoms
Socio-Demography | Pre-assessment (-2 weeks), Baseline (0 weeks)
  Self-reported height, weight, education, work-situation, family-situation, and socio-economic status
Emotional Distress subscale of the 92-item version of the Symptom Checklist (SCL-92_DIST) | During treatment (weeks 3, 6, 9)
  Self-reported Emotional Distress symptoms
European Quality of Life 5-dimensions (EQ-5D-5L) | Baseline (0 weeks), after treatment (14 weeks) at 3-month follow up (26 weeks) and at 12-month follow up (62 weeks).
  Self-reported quality of life measure

OTHER OUTCOMES:
Automatic log data | Data is logged throughout entire treatment period. This data will be collected from baseline (0 weeks) and throughout the treatment period (week 14).
  The follow variables are logged variables: The follow variables are logged variables: Time spent in program; Modules and pages; Number of logins; Number of completed modules; Activities engaged with (e.g. exercises interacted with); Textual content of all text boxes.
End-of-module evaluation | Not time specific, but collected throughout the usage-period, when users complete a module. This data will be collected from baseline (0 weeks) and throughout the treatment period (week 14)
  Self-reported single item questions regarding the experience of working within each module
Assessing medical doctor evaluation | Immediately following assessment (-2 weeks), after 3 month follow-up assessment (30 weeks)
  Medical doctor responsible for assessment and inclusion will note to which degree patients live up to inclusion criteria, and make an assessment of clinical characteristics and barriers to treatment.
Therapist evaluation of phone consultations | During the entire treatment period (from week 0 to week 14)
  Date and theme of phone consultations
Therapist rated time usage, motivation and treatment barriers for patient | After treatment (14 weeks)
  Patients motivation and barriers to treatment is assessed after ended treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Frostholm, Ph.D., Principal Investigator — Aarhus Universityhospital
Locations (1):
- Department of Functional Disorders, Aarhus C, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schroder A, Rehfeld E, Ornbol E, Sharpe M, Licht RW, Fink P. Cognitive-behavioural group treatment for a range of functional somatic syndromes: randomised trial. Br J Psychiatry. 2012 Jun;200(6):499-507. doi: 10.1192/bjp.bp.111.098681. Epub 2012 Apr 26. PMID 22539780
- [Background] Fjorback LO, Arendt M, Ornbol E, Walach H, Rehfeld E, Schroder A, Fink P. Mindfulness therapy for somatization disorder and functional somatic syndromes: randomized trial with one-year follow-up. J Psychosom Res. 2013 Jan;74(1):31-40. doi: 10.1016/j.jpsychores.2012.09.006. Epub 2012 Oct 1. PMID 23272986
- [Background] Pedersen HF, Agger JL, Frostholm L, Jensen JS, Ornbol E, Fink P, Schroder A. Acceptance and Commitment group Therapy for patients with multiple functional somatic syndromes: a three-armed trial comparing ACT in a brief and extended version with enhanced care - CORRIGENDUM. Psychol Med. 2018 Dec;48(16):2804. doi: 10.1017/S0033291718002799. Epub 2018 Sep 11. No abstract available. PMID 30203729
- [Background] Frolund Pedersen H, Holsting A, Frostholm L, Rask C, Jensen JS, Hoeg MD, Schroder A. "Understand your illness and your needs": Assessment-informed patient education for people with multiple functional somatic syndromes. Patient Educ Couns. 2019 Sep;102(9):1662-1671. doi: 10.1016/j.pec.2019.04.016. Epub 2019 Apr 17. PMID 31023608
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681